CLINICAL TRIAL: NCT05841277
Title: Pharmacokinetics of LY3819469 Following Subcutaneous Dose in Participants With Renal Impairment Compared With Participants With Normal Renal Function
Brief Title: A Study of LY3819469 in Participants With Impaired and Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18731; J3L-MC-EZED (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3819469 (Control) (Experimental): LY3819469 administered subcutaneously (SC) to participants with normal renal function
  Interventions: Drug: LY3819469
- LY3819469 (Severe Renal Impairment) (Experimental): LY3819469 administered SC to participants with severe renal impairment
  Interventions: Drug: LY3819469
- LY3819469 (End-Stage Renal Disease) (Experimental): LY3819469 administered SC to participants with end-stage renal disease (ESRD)
  Interventions: Drug: LY3819469

INTERVENTIONS:
Drug: LY3819469 — Administered SC.

SUMMARY:
The main purpose of this study is to assess the amount of study drug (LY3819469) that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment compared to participants with normal renal function. The safety and tolerability of LY3819469 will also be evaluated in these participants. The study will last up to 17 weeks including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index within the range 19.0 to 42.0 kilograms per meter squared (kg/m²)
* Men who agree to use highly effective or effective methods of contraception and women not of childbearing potential (WNOCBP) may participate in this trial

Participants with Normal Renal Function:

* Have estimated glomerular filtration rate (eGFR) determined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) greater than or equal to 90 milliliter per minute (mL/min)

Participants with Renal Impairment:

* Severe renal impairment: Have eGFR determined by CKD-EPI of less than 30 mL/min and not requiring dialysis
* ESRD: Participants who have been on a stable hemodialysis schedule for at least 3 months prior to planned dosing

Exclusion Criteria:

* Have a history or presence of an underlying disease, or surgical, physical, medical, or psychiatric condition
* Have any abnormality in the 12-lead electrocardiogram (ECG)
* Hemoglobin less than 8 grams per deciliter (g/dL) and clinically significant anemia symptoms
* Have known allergies to LY3819469, related compounds or any components of the formulation, or a history of significant atopy
* Have participated in any Lp(a) siRNA therapeutic clinical trial within the last 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to last time point (AUC0-tlast) of LY3819469 | Predose up to 85 days postdose
  PK: AUC0-tlast of LY3819469
PK: Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3819469 | Predose up to 85 days postdose
  PK: AUC0-∞ of LY3819469
PK: Maximum observed concentration (Cmax) of LY3819469 | Predose up to 85 days postdose
  PK: Cmax of LY3819469

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Floridian Clinical Research, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - Nucleus Networks, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No